CLINICAL TRIAL: NCT01390142
Title: Remote Ischemic Preconditioning Combined to Local Ischemic Postconditioning in Acute Myocardial Infarction (RIRE-1)
Brief Title: Remote Ischemic Preconditioning Combined to Local Ischemic Postconditioning in Acute Myocardial Infarction
Acronym: RIRE-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Fédération Française de Cardiologie (Other); Société Française de Cardiologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC 2011-06
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-10

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

ARMS (3):
- Control (Experimental)
  Interventions: Procedure: Control
- RIPer (Active Comparator): Remote ischemic preconditioning
  Interventions: Procedure: RIPer
- RIPer + IPost (Active Comparator): Remote ischemic preconditioning and Local ischemic postconditioning
  Interventions: Procedure: RIPer + IPost

INTERVENTIONS:
Procedure: Control — Deflated blood pressure cuff placed on upper arm for 30min
  Arms: Control
Procedure: RIPer — Blood pressure cuff placed on upper arm and inflated to 200 mmHg for 5 min and then deflated for 5 min. This cycle is initiated as soon as possible after patient admission in the cathlab and repeated 3 times in total.
  Arms: RIPer
Procedure: RIPer + IPost — Blood pressure cuff placed on upper arm and inflated to 200 mmHg for 5 min and then deflated for 5 min. This cycle is initiated as soon as possible after patient admission in the cathlab and repeated 3 times in total. Within the first minute of re-established coronary flow by primo-stenting, the same balloon is re-inflated for 1 min and then deflated for 1min. This procedure of balloon inflation/deflation is repeated 4 times in total.
  Arms: RIPer + IPost

SUMMARY:
RIRE-1 is a randomized, open-label with blinded end-point study that will test the hypothesis that remote ischemic preconditioning initiated at the time of the admission in the cathlab reduces infarct size in ST-segment elevation myocardial infarction (STEMI) patients treated with percutaneous coronary intervention (PCI). Furthermore, it will determine whether a combined approach remote ischemic preconditioning and local ischemic postconditioning can further reduce infarct size. Infarct size will be determined by cardiac magnetic resonance imaging at 3-month follow-up and with 72 hours area under curve of CK-MB.

DETAILED DESCRIPTION:
In the management of STEMI, prompt reperfusion of the jeopardized myocardium is the most effective way to limit infarct size, which is a major determinant of morbidity and mortality. However, restoration of blood flow may paradoxically have deleterious consequences and lead to lethal myocardial ischemia-reperfusion injury. Local ischemic postconditioning (IPost) and remote ischemic preconditioning (RIPer) are promising methods to decrease ischemia-reperfusion injury.

The hypothesis tested in this research proposal is that RIPer initiated at the time of the admission in the cathlab reduces infarct size in STEMI patients treated with PCI. Furthermore, the investigators will determine whether a combined approach RIPer + IPost can further reduce infarct size.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* ST-Segment elevation myocardial infarction <6h
* Written informed consent

Exclusion Criteria:

* Previous Q-wave myocardial infarction or previous coronary artery bypass graft
* Cardiogenic shock
* Cardiac arrest resuscitated before angioplasty
* Infarct related artery : circumflex coronary artery, right coronary artery after segment 3, left main, diagonal and marginal branches, and all coronary artery with jeopardized myocardium estimated too small.
* TIMI 2 or 3 before angioplasty
* Collateral branches Rentrop >1
* TIMI 0 or 1 flow grade after PCI
* Any contraindications to magnetic resonance imaging
* Allergy to gadolinium
* Patient refusal / patient not having provided written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Infarct size | 3 months
  Infarct size as assessed by 72 hours area under curve serum CK-MB and cardiac magnetic resonance imaging at 3-month follow-up

SECONDARY OUTCOMES:
Microvascular obstruction | 5 days
  Microvascular obstruction as assessed by cardiac magnetic resonance imaging at 5-day follow-up
Left ventricular remodeling | 3 months
  Left ventricular remodeling as assessed by cardiac magnetic resonance imaging at 5-day and 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Prunier, MD, PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- CHU Angers - Service de Cardiologie, Angers, France